CLINICAL TRIAL: NCT07222371
Title: An Open-label, Single Center, Single Participant Study of an Experimental Antisense Oligonucleotide Treatment for TUBB4A-related Leukodystrophy
Acronym: ASOTUBB4A
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Olivia Kim-McManus, Professor, Neurosiences, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 812067
Record Dates: First submitted 2025-10-27; First posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: Genetic Disease; TUBB4A-Related Leukodystrophy
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open label (Experimental)
  Interventions: Drug: nL-TUBB4-001

INTERVENTIONS:
Drug: nL-TUBB4-001 — Personalized antisense oligonucleotide

SUMMARY:
This current study is aimed for the treatment of an individual participant with a form of TUBB4A-related leukodystrophy with hypomyelination.

DETAILED DESCRIPTION:
The study is an investigational interventional drug created for the study subject's specific pathogenic genetic mutation.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent/assent provided by the participant (when appropriate), and/or participant's parent(s) or legally authorized representative(s).
* Ability to travel to the study site and adhere to study-related follow-up examinations and/or procedures and provide access to participant's medical records.
* Clinical phenotype and neuroimaging consistent with a diagnosis of TUBB4A-related leukodystrophy
* Documented genetic mutation in TUBB4A

Exclusion Criteria:

* Participant has any known contraindication to or unwillingness to undergo lumbar puncture
* Use of investigational medication within 5 half-lives of the drug at enrollment
* Participant has any condition that in the opinion of the Site Investigator, would ultimately prevent the completion of study procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2025-09-19 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Dystonia and gross motor function as measured by Barry Albright Dystonia Scale (BAD) | baseline to 12 and 24 months
  The Barry Albright Dystonia Scale (BAD) is a clinical tool designed to evaluate the severity of dystonia in children. This scale assesses dystonia in eight different body regions including the eyes, mouth, neck, trunk, and each of the four limbs. Each region is scored on a severity scale from 0 (no dystonia) to 4 (severe dystonia), allow for quantification of the overall dystonia as well as distribution of dystonic movements across the body. The BAD will be performed at each study timepoint as specified by SoA by the same trained and qualified administrator.
Dystonia and gross motor function as measured by Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS) | baseline to 12 and 24 months
  The Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS) assesses the severity of dystonia as well as its impact on daily life. It consists of two main components: the Movement Scale, which scores dystonia in various body regions such as the eyes, mouth, neck, trunk, and limbs on a scale from 0 (no dystonia) to 4 (severe dystonia), and the Disability Scale, which evaluates the impact of dystonia on daily activities (e.g., feeding, hygiene, dressing, etc.).
Dystonia and gross motor function as measured by Gross Motor Function Measure-88 (GMFM-88) | baseline to 12 and 24 months
  The Gross Motor Function Measure-88 (GMFM-88) evaluates changes in gross motor function in children with conditions that affect gross motor abilities. Motor function is assessed through 88 tasks across five dimensions: lying and rolling, sitting, crawling, and kneeling, standing, and walking, running, and jumping. Each item is scored on a four-point ordinal scale based on observed performance, providing quantification of gross motor function and the ability to track progress or regression over time.
Dystonia and gross motor function as measured by Vineland Adaptive Behavior Scales | baseline to 12 and 24 months
  The Vineland Adaptive Behavior Scales, Third Edition (Vineland-3), is a standardized, validated, and reliable assessment tool designed to measure the adaptive behavior of individuals from birth through adulthood. The Vineland-3 Motor Skills domain evaluates gross and fine motor abilities in individuals from birth to age 9, offering insights into coordination, balance, mobility, and dexterity. The raw scores are converted to standard scores and growth scale value scores, with higher scores indicating better adaptive functioning.

SECONDARY OUTCOMES:
Communication, behavioral and cognitive skills measured by The Vineland Adaptive Behavior Scales | baseline to 12 and 24 months
  The Vineland Adaptive Behavior Scales, Third Edition (Vineland-3), is a standardized, validated, and reliable assessment tool designed to measure the adaptive behavior of individuals from birth through adulthood. The Vineland-3 Motor Skills domain evaluates gross and fine motor abilities in individuals from birth to age 9, offering insights into coordination, balance, mobility, and dexterity. The raw scores are converted to standard scores and growth scale value scores, with higher scores indicating better adaptive functioning.
Communication, behavioral and cognitive skills measured bythe Bayley Scales of Infant and Toddler Development 4th Edition (BSID-4) | baseline to 12 and 24 months
  The Bayley Scales of Infant and Toddler Development is a standardized, validated, and reliable assessment tool for evaluating developmental functioning in infants and toddlers. Its Motor Skills domain evaluates gross and fine motor abilities, including coordination, balance, and movement. The raw scores are converted to standard scores and growth scale value scores, with higher scores indicating better motor development.
Quality of life as measured by PedsQL Family Impact Module | baseline to 6-, 12-, 18-, and 24-months
  The Pediatric Quality of Life Inventory (PedsQL) Family Impact Module is a multidimensional instrument developed to assess the impact of chronic medical conditions on the health-related quality of life of parents and family functioning. This module measures parents' self-reported physical, emotional, social, and cognitive functioning, communication, and worry. The PedsQL Family Impact Module has shown reliability and validity in families with children with complex chronic health conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Rady Children's Hospital San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No